CLINICAL TRIAL: NCT05074420
Title: A Multicenter, Open-Label, Pharmacokinetic and Safety Study of Baricitinib in Pediatric Patients From 1 Year to Less Than 18 Years Old Hospitalized With COVID-19
Brief Title: A Study of Baricitinib (LY3009104) in Children With COVID-19
Acronym: COV-BARRIER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to an inability to enroll participants.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18253; I4V-MC-KHAB (Other: Eli Lilly and Company); 2021-001338-21 (EudraCT Number)
Record Dates: First submitted 2021-10-08; First posted 2021-10-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Covid19; Corona Virus Infection
Keywords: coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Baricitinib (Experimental): Baricitinib given orally to participants daily
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Given Orally
  Other Names: LY3009104

SUMMARY:
The purpose for this study is to determine if the study drug baricitinib is effective and safe in hospitalized pediatric participants with Coronavirus disease 2019 (COVID -19) and to confirm the dose.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with coronavirus (SARS-CoV-2) infection.
* Male or female participants from 1 to <18 years of age.
* Requires supplemental oxygen and have chest imaging findings to confirm respiratory disease due to COVID-19 within 72 hours of study entry and enrollment.
* Supplemental oxygen including but not limited to: nasal cannula, mask, high flow devices, CPAP/BiPAP, invasive mechanical ventilation as well as ECMO.

Exclusion Criteria:

* Are receiving biologic treatments (such as Tumor Necrosis Factor [TNF] inhibitors, interleukin inhibitors, T-cell or B-cell targeted therapies, interferon, or Janus kinase (JAK) inhibitors); or are receiving other immunosuppressants such that, in the opinion of the investigator, participating in the study would put the participant at an unacceptable risk of immunosuppression.

Note: A washout period is required prior to screening.

* Are receiving strong inhibitors of Organic Anion Transporter 3 (OAT3) (such as probenecid) that cannot be discontinued at study entry.
* Have diagnosis of current active tuberculosis (TB) or, if known, latent TB treated for less than 4 weeks with appropriate anti-tuberculosis therapy per local guidelines (by history only, no screening tests required).
* Suspected serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking investigational product.
* Have received any live vaccine within 4 weeks before screening, or intend to receive a live vaccine during the study. Note: Use of non-live (inactivated) vaccinations are allowed for all participants.
* Require invasive mechanical ventilation, including extracorporeal membrane oxygenation (ECMO) at study entry.
* Current diagnosis of active malignancy that, in the opinion of the investigator, could constitute a risk when taking investigational product.
* Have a history of venous thromboembolism (VTE) (deep vein thrombosis [DVT] and/or pulmonary embolism [PE]) or considered high risk of VTE (DVT/PE).
* Anticipated discharge from the hospital, or transfer to another hospital (or another unit), which is not a study site within 72 hours after study entry.
* Have neutropenia (absolute neutrophil count <1000 cells/microliters).
* Have lymphopenia (absolute lymphocyte count <200 cells/microliters).
* Have alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 times AAULN.
* Estimated glomerular filtration rate (eGFR) (Modification of Diet in Renal Disease [MDRD]) <40 milliliter/minute/1.73 meters squared.
* Have a known hypersensitivity to baricitinib or any of its excipients.
* Are currently enrolled in any other clinical study involving an investigation product or any other type of medical research judged not to be scientifically or medically compatible with this study. Note: The participant should not be enrolled (started) in another clinical trial for the treatment of COVID-19 or SARS CoV-2 through Day 28.
* Are pregnant, or intend to become pregnant or breastfeed during the study.
* Are, in the opinion of the investigator or sponsor, at risk of immunosuppression or otherwise unsuitable for inclusion in the study.
* Are using or will use extracorporeal blood purification (EBP) device to remove proinflammatory cytokines from the blood such as a cytokine absorption or filtering device, for example, CytoSorb®.
* Are, in the opinion of the investigator, unlikely to survive for at least 48 hours after screening.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under Concentration Curve (AUC) of Baricitinib | Day 1 and Day 4
  PK: AUC of Baricitinib in pediatric participants with COVID-19
PK: Maximum Concentration (Cmax) of Baricitinib | Day 1 and Day 4
  PK: Cmax of Baricitinib in pediatric participants with COVID-19

SECONDARY OUTCOMES:
Percentage of Participants Who Require Noninvasive Ventilation/high-flow oxygen or Invasive Mechanical Ventilation (including extracorporeal membrane oxygenation [ECMO]) | Day 1 to Day 28
  Percentage of participants who require noninvasive ventilation/high-flow oxygen or invasive mechanical ventilation (including ECMO)
Percentage of Participants Who Die or Require Non-Invasive Ventilation/High-Flow Oxygen or Invasive Mechanical Ventilation (including ECMO) | Day 1 to Day 28
  Percentage of Participants who Die or Require Non-Invasive Ventilation/High-Flow Oxygen or Invasive Mechanical Ventilation (including ECMO)
Percentage of Participants with at Least 1-Point Improvement on National Institute of Allergy and Infectious Diseases Ordinal Scale (NIAID-OS) or Live Discharge from Hospital | Day 4, Day 7, Day 10, Day 14, and Day 28
  Percentage of Participants with at Least 1-Point Improvement on NIAID-OS or Live Discharge from Hospital. The NIAID-OS scale ranges from 1 - 8 (worse outcome).
Number of Ventilator-Free Days | Day 1 to Day 28
  Number of Ventilator-Free Days
Time to Recovery | Day 1 to Day 28
  Recovery assessed by the NIAID-OS
Overall improvement on the NIAID-OS | Day 4, Day 7, Day 10, Day 14, and Day 28
  Overall improvement on the NIAID-OS
Duration of Hospitalization | Day 1 to Day 28
  Duration of Hospitalization
All-Cause Mortality | Day 1 to Day 28 and Day 60
  All-Cause Mortality
Duration of Stay in the Intensive Care Unit (ICU) in Days | Day 1 to Day 28
  Duration of Stay in the ICU in Days

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (3):
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Children's Hospital of Michigan, Detroit, Michigan
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- Brazil (5):
  - Centro de Pesquisa Sao Lucas, Campinas
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - CECIP - Centro de Estudos do Interior Paulista, Jaú
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Pesquisare Saude, Santo André
- Mexico (2):
  - Instituto Nacional de Pediatria, Mexico City
  - Hospital Infantil de Mexico Federico Gomez, Mexico City
- Spain (4):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario de Araba (HUA)- Hospital Txagorritxu, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Baricitinib (LY3009104) in Children With COVID-19 (COV-BARRIER-PEDS) — https://trials.lilly.com/en-US/trial/306960